CLINICAL TRIAL: NCT03392168
Title: A Phase 1/2a Single Dose and 28-day Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety, Pharmacokinetics and Efficacy of ARQ-151 Cream 0.5% and 0.15% in Adults With Mild to Moderate Chronic Plaque Psoriasis
Brief Title: Safety, Pharmacokinetics and Efficacy of ARQ-151 Cream in Adults With Mild to Moderate Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARQ-151-101
Record Dates: First submitted 2017-12-29; First posted 2018-01-05 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Psoriasis
Keywords: Psoriasis; Plaque Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohort 1 was open label. Cohort 2 was double blind.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 - ARQ-151 cream 0.5% (Experimental): Single-dose application of ARQ-151 cream 0.5% to 25 cm^2 of psoriatic plaque(s)
  Interventions: Drug: ARQ-151 cream 0.5%
- Cohort 2 - ARQ-151 cream 0.5% (Experimental): ARQ-151 cream 0.5% applied daily for 28 days to all psoriatic plaques, not exceeding an application area of 5% BSA
  Interventions: Drug: ARQ-151 cream 0.5%
- Cohort 2 - ARQ-151 cream 0.15% (Experimental): ARQ-151 cream 0.15% applied daily for 28 days to all psoriatic plaques, not exceeding an application area of 5% BSA
  Interventions: Drug: ARQ-151 cream 0.15%
- Cohort 2 - ARQ-151 vehicle cream (Placebo Comparator): Vehicle cream applied daily for 28 days to all psoriatic plaques, not exceeding an application area of 5% BSA
  Interventions: Drug: ARQ-151 vehicle cream

INTERVENTIONS:
Drug: ARQ-151 cream 0.5% — 0.5% active concentration
  Arms: Cohort 1 - ARQ-151 cream 0.5%; Cohort 2 - ARQ-151 cream 0.5%
Drug: ARQ-151 cream 0.15% — 0.15% active concentration
  Arms: Cohort 2 - ARQ-151 cream 0.15%
Drug: ARQ-151 vehicle cream — Vehicle cream
  Arms: Cohort 2 - ARQ-151 vehicle cream

SUMMARY:
This study assessed the safety and pharmacokinetics (PK) of a single dose application of ARQ-151 cream 0.5% to 25 cm^2 of psoriatic plaque(s) (Cohort 1). The study also assessed the safety, PK and efficacy of ARQ-151 cream 0.5% vs vehicle and ARQ-151 cream 0.15% vs vehicle applied once a day for 28 days to individuals with 0.5% to 5.0% body surface area (BSA) of chronic plaque psoriasis (Cohort 2).

DETAILED DESCRIPTION:
There were 2 cohorts of participants. Cohort 1 was a single dose study of ARQ-151 0.5% cream applied to 25 cm^2 of psoriatic plaque(s) in 8 psoriasis participants. Cohort 2 was a parallel group, double blind, vehicle controlled study in which ARQ-151 cream 0.5%, ARQ-151 cream 0.15% or vehicle cream was applied once a day for 28 days to participants with between 0.5% to 5.0% BSA of chronic plaque psoriasis. Participants were adult (≥18 years old) males or females with chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female participants aged ≥18 years.
* In Cohort 1, participants must have at least 25 cm^2 of chronic plaque psoriasis (excluding the face, scalp, intertriginous areas, palms and soles).
* In Cohort 2, participants must have 0.5% to 5.0% of total BSA of chronic plaque psoriasis and at least one target plaque, of at least 9 cm^2 in size with a TPSS ≥4 (excluding the face, scalp, intertriginous areas, palms and soles).
* Women of childbearing potential must have a negative urine pregnancy test at Screening and agree to use birth control throughout the trial.
* In good health as judged by the Investigator, based on medical history, physical examination, 12-lead electrocardiogram (ECG), serum chemistry labs, hematology values, and urinalysis.
* Participants agree not to have prolonged sun exposure during the course of the study. Tanning bed use is not allowed.
* Participants are competent to sign and give informed consent and considered reliable and capable of adhering to the Protocol and visit schedule.

Exclusion Criteria:

* Participants with non-plaque forms of psoriasis (erythrodermic, guttate, pustular or palmo-plantar psoriasis) or with drug-induced psoriasis.
* Evidence of skin conditions other than psoriasis that would interfere with evaluation of the effect of the study medication.
* Pregnant or lactating women or women planning to become pregnant during the study and / or within 28 days following the last dose of study medication.
* Known allergies to excipients in ARQ-151 cream.
* Participants who cannot discontinue the use of strong P-450 cytochrome inducers or inhibitors for two weeks prior to the baseline visit and during the study period.
* Participants who are unwilling to refrain from using a tanning bed for 2 weeks before and during the study.
* Participants who cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis.
* Participants with a history of chronic alcohol or drug abuse in past 6 months.
* History of and/or concurrent condition of serious hypersensitivity (anaphylactic shock or anaphylactoid reaction) to phosphodiesterase type 4 (PDE-4) inhibitors.
* Current or a history of cancer within 5 years with the exception of fully excised skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix.
* Participants with active infection that requires oral or intravenous administration of antibiotics, antifungal or antiviral agents.
* Participants who are unable to communicate, read or understand language, or who display another condition which makes them unsuitable for clinical study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, M.D., Study Director — Arcutis Biotherapeutics, Inc.
Locations (8):
- Mosaic Dermatology, Santa Monica, California, United States
- Canada (7):
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Lynderm Research Inc., Markham, Ontario
  - Research by ICLS, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thurston AW Jr, Osborne DW, Snyder S, Higham RC, Burnett P, Berk DR. Pharmacokinetics of Roflumilast Cream in Chronic Plaque Psoriasis: Data from Phase I to Phase III Studies. Am J Clin Dermatol. 2023 Mar;24(2):315-324. doi: 10.1007/s40257-022-00741-9. Epub 2022 Nov 24. PMID 36422852
- [Derived] Papp KA, Gooderham M, Droege M, Merritt C, Osborne DW, Berk DR, Thurston AW, Smith VH, Welgus H. Roflumilast Cream Improves Signs and Symptoms of Plaque Psoriasis: Results from a Phase 1/2a Randomized, Controlled Study. J Drugs Dermatol. 2020 Aug 1;19(8):734-740. doi: 10.36849/JDD.2020.5370. PMID 32845114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 7 centers in Canada and 1 center in the United States (US). There was a total of 91 unique participants; 6 participants who completed Cohort 1 also participated in Cohort 2, with 2 per treatment group.
Period: Period 1: Cohort 1
Arm/Group | Cohort 1 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream
Started | 8 | 0 | 0 | 0
Completed | 8 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Period 2: Cohort 2
Arm/Group | Cohort 1 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream
Started | 0 | 30 (Includes 2 participants from Cohort 1) | 28 (Includes 2 participants from Cohort 1) | 31 (Includes 2 participants from Cohort 1)
Completed | 0 | 28 | 27 | 30
Not Completed | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics for Cohort 2 arms are shown for participants who were not in Cohort 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream | Total
Number analyzed (Participants) | 8 | 28 | 26 | 29 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.6 (16.92) | 50.8 (15.76) | 54.8 (13.50) | 47.0 (13.97) | 50.80 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 7 | 12 | 38
  Male | 1 | 16 | 19 | 17 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 27 | 26 | 29 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 2 | 0 | 4
  White | 8 | 23 | 22 | 20 | 73
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 4 Week Target Plaque Severity Score x Target Plaque Area in Cohort 2
Description: Difference in least squares mean percent change from baseline at Week 4 in the product of target plaque severity score (TPSS) x target plaque area (TPA) between each dose concentration level of ARQ-151 cream and vehicle using mixed model repeated measures (MMRM) analysis with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects and baseline TPSS x TPA score as a covariate. For TPSS, all target lesions were scored individually for signs of induration, scaling, and erythema using a 5-point severity scale: 0 = none; 1 = mild; 2 = moderate; 3 = severe; 4 = very severe. TPA (cm^2) was determined by multiplying the longest diameter (cm) of the target plaque by the widest perpendicular diameter (cm) (perpendicular to the longest diameter of the target plaque). A negative percent change indicates improvement.
Time Frame: Baseline and Week 4
Population: The modified intent-to-treat (mITT) population included all participants who were in the safety population for Cohort 2 with at least 1 postbaseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream
Number analyzed (Participants) | 28 | 27 | 30
Percent change | -66.6 (7.27) | -66.0 (7.61) | -38.1 (7.34)
Statistical Analysis 1: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; LS mean difference from vehicle; Estimates for LS means and accompanying 95% confidence intervals and P values are from a mixed model for repeated measures (MMRM) with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects, and baseline value as a covariate; Test type: Superiority; p = 0.0007, Mixed Models Analysis; Least squares mean difference = -28.5, 95% CI 2-sided [-44.6 to -12.4]
Statistical Analysis 2: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0011, Mixed Models Analysis; Least squares mean difference = -27.8, 95% CI 2-sided [-44.2 to -11.5]

2. Secondary Outcome: Percent Change From Baseline in 1, 2, 3 Week Target Plaque Severity Score x Target Plaque Area in Cohort 2
Description: Difference in least squares mean percent change from baseline at Weeks 1, 2 and 3 in target plaque severity score (TPSS) x target plaque area (TPA) between each dose concentration level of ARQ-151 cream and vehicle using mixed model repeated measures (MMRM) analysis with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects and baseline TPSS x TPA score as a covariate. For TPSS, all target lesions were scored individually for signs of induration, scaling, and erythema using a 5-point severity scale: 0 = none; 1 = mild; 2 = moderate; 3 = severe; 4 = very severe. TPA (cm^2) was determined by multiplying the longest diameter (cm) of the target plaque by the widest perpendicular diameter (cm) (perpendicular to the longest diameter of the target plaque). A negative percent change indicates improvement.
Time Frame: Baseline and Weeks 1, 2 and 3
Population: The mITT population included all participants who were in the safety population for Cohort 2 with at least 1 postbaseline efficacy evaluation.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream
Number analyzed (Participants) | 30 | 27 | 31
Percent change
  Week 1 | -34.7 (5.79) | -36.4 (6.16) | -31.5 (5.99)
  Week 2: number analyzed (Participants) | 28 | 27 | 30
  Week 2 | -48.7 (6.40) | -50.1 (6.75) | -30.4 (6.55)
  Week 3: number analyzed (Participants) | 28 | 27 | 30
  Week 3 | -61.5 (6.69) | -55.6 (7.03) | -32.6 (6.81)
Statistical Analysis 1: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; At Week 1; LS mean difference from vehicle; Estimates for LS means and accompanying 95% confidence intervals and P values are from a mixed model for repeated measures (MMRM) with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects, and baseline value as a covariate; Test type: Superiority; p = 0.5493, Mixed Models Analysis; Least squares mean difference = -3.2, 95% CI 2-sided [-13.7 to 7.3]
Statistical Analysis 2: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3650, Mixed Models Analysis; Least squares mean difference = -4.9, 95% CI 2-sided [-15.7 to 5.9]
Statistical Analysis 3: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; At Week 2; LS mean difference from vehicle; Estimates for LS means and accompanying 95% confidence intervals and P values are from a mixed model for repeated measures (MMRM) with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects, and baseline value as a covariate; Test type: Superiority; p = 0.0064, Mixed Models Analysis; Least squares mean difference = -18.3, 95% CI 2-sided [-31.3 to -5.3]
Statistical Analysis 4: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.0039, Mixed Models Analysis; Least squares mean difference = -19.8, 95% CI 2-sided [-33.0 to -6.5]
Statistical Analysis 5: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; At Week 3; LS mean difference from vehicle; Estimates for LS means and accompanying 95% confidence intervals and P values are from a mixed model for repeated measures (MMRM) with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects, and baseline value as a covariate; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Least squares mean difference = -28.9, 95% CI 2-sided [-42.9 to -14.8]
Statistical Analysis 6: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.0019, Mixed Models Analysis; Least squares mean difference = -23.0, 95% CI 2-sided [-37.3 to -8.7]

3. Secondary Outcome: Percent Change From Baseline in Total Plaque Severity Score in Cohort 2
Description: Difference in least squares mean percent change from baseline at Weeks 1, 2, 3 and 4 in total plaque severity score (TPSS) between each dose concentration level of ARQ-151 cream and vehicle using mixed model repeated measures (MMRM) analysis with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects and baseline TPSS score as a covariate. For TPSS, all target lesions were scored individually for signs of induration, scaling, and erythema using a 5-point severity scale: 0 = none; 1 = mild; 2 = moderate; 3 = severe; 4 = very severe. A negative percent change indicates improvement.
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream
Number analyzed (Participants) | 30 | 27 | 31
Percent change
  Week 1 | -30.5 (4.96) | -34.3 (5.20) | -26.2 (5.16)
  Week 2: number analyzed (Participants) | 28 | 27 | 30
  Week 2 | -41.9 (5.01) | -45.6 (5.22) | -26.4 (5.19)
  Week 3: number analyzed (Participants) | 28 | 27 | 30
  Week 3 | -51.5 (5.46) | -52.0 (5.63) | -30.1 (5.56)
  Week 4: number analyzed (Participants) | 28 | 27 | 30
  Week 4 | -55.1 (5.41) | -58.2 (5.56) | -36.5 (5.50)
Statistical Analysis 1: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3626, Mixed Models Analysis; Least squares mean difference = -4.3, 95% CI 2-sided [-13.6 to 5.0]
Statistical Analysis 2: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1011, Mixed Models Analysis; Least squares mean difference = -8.1, 95% CI 2-sided [-17.8 to 1.6]
Statistical Analysis 3: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.0017, Mixed Models Analysis; Least squares mean difference = -15.5, 95% CI 2-sided [-25.1 to -6.0]
Statistical Analysis 4: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Least squares mean difference = -19.3, 95% CI 2-sided [-29.1 to -9.4]
Statistical Analysis 5: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Least squares mean difference = -21.3, 95% CI 2-sided [-32.4 to -10.2]
Statistical Analysis 6: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Least squares mean difference = -21.8, 95% CI 2-sided [-33.2 to -10.4]
Statistical Analysis 7: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; At Week 4; LS mean difference from vehicle; Estimates for LS means and accompanying 95% confidence intervals and P values are from a mixed model for repeated measures (MMRM) with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects, and baseline value as a covariate; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Least squares mean difference = -18.7, 95% CI 2-sided [-29.5 to -7.8]
Statistical Analysis 8: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Least squares mean difference = -21.8, 95% CI 2-sided [-32.9 to -10.6]

4. Secondary Outcome: Percent Change From Baseline in Target Plaque Area in Cohort 2
Description: Difference in least squares mean percent change from baseline at Weeks 1, 2, 3, and 4 in target plaque area (TPA) between each dose concentration level of ARQ-151 cream and vehicle using mixed model repeated measures (MMRM) analysis with center within country, treatment, study visit, and treatment-by-study visit interaction as fixed effects and baseline TPA score as a covariate. Target plaque area (cm^2) was determined by multiplying the longest diameter (cm) of the target plaque by the widest perpendicular diameter (cm) (perpendicular to the longest diameter of the target plaque). A negative percent change indicates improvement.
Time Frame: Baseline and Weeks 1, 2, 3, and 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream
Number analyzed (Participants) | 30 | 27 | 31
Percent change
  Week 1 | -9.15 (2.981) | -8.22 (3.198) | -11.82 (3.089)
  Week 2: number analyzed (Participants) | 28 | 27 | 30
  Week 2 | -14.95 (4.211) | -16.19 (4.407) | -10.37 (4.225)
  Week 3: number analyzed (Participants) | 28 | 27 | 30
  Week 3 | -22.63 (4.666) | -17.00 (4.844) | -9.95 (4.636)
  Week 4: number analyzed (Participants) | 28 | 27 | 30
  Week 4 | -31.87 (6.014) | -28.28 (6.228) | -11.61 (5.938)
Statistical Analysis 1: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3209, Mixed Models Analysis; Least squares mean difference = 2.67, 95% CI 2-sided [-2.65 to 7.99]
Statistical Analysis 2: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1947, Mixed Models Analysis; Least squares mean difference = 3.60, 95% CI 2-sided [-1.88 to 9.08]
Statistical Analysis 3: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.3561, Mixed Models Analysis; Least squares mean difference = -4.58, 95% CI 2-sided [-14.40 to 5.24]
Statistical Analysis 4: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.2490, Mixed Models Analysis; Least squares mean difference = -5.82, 95% CI 2-sided [-15.79 to 4.16]
Statistical Analysis 5: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.0276, Mixed Models Analysis; Least squares mean difference = -12.68, 95% CI 2-sided [-23.992 to -1.44]
Statistical Analysis 6: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 2, analysis 5]; Test type: Superiority; p = 0.2223, Mixed Models Analysis; Least squares mean difference = -7.04, 95% CI 2-sided [-18.44 to 4.36]
Statistical Analysis 7: Comparison: Cohort 2 - ARQ-151 Cream 0.5% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0108, Mixed Models Analysis; Least squares mean difference = -20.27, 95% CI 2-sided [-35.72 to -4.82]
Statistical Analysis 8: Comparison: Cohort 2 - ARQ-151 Cream 0.15% vs Cohort 2 - ARQ-151 Vehicle Cream; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p = 0.0372, Mixed Models Analysis; Least squares mean difference = -16.67, 95% CI 2-sided [-32.34 to -1.01]

ADVERSE EVENTS:
Time Frame: Up to approximately 5 months
Description: A treatment-emergent adverse event is an event that is temporally associated with administration of study product; events meeting this definition are those with a start date during or after administration of the first dose of study drug through the telephone follow-up in each cohort.
Arm/Group | Cohort 1 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.5% | Cohort 2 - ARQ-151 Cream 0.15% | Cohort 2 - ARQ-151 Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/30 | 0/28 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/30 | 0/28 | 0/31
Other Adverse Events (participants affected / at risk) | 1/8 | 9/30 | 5/28 | 11/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - ARQ-151 Cream 0.5% (N=8) | Cohort 2 - ARQ-151 Cream 0.5% (N=30) | Cohort 2 - ARQ-151 Cream 0.15% (N=28) | Cohort 2 - ARQ-151 Vehicle Cream (N=31)
Application site erythema (General disorders) | 0 (0) | 4 (4) | 1 (1) | 4 (4)
Application site pain (General disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Candiduria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT03392168/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT03392168/SAP_001.pdf